CLINICAL TRIAL: NCT01763762
Title: A Comparison of the Efficacy of Electrical Pudendal Nerve Stimulation to Pelvic Floor Muscle Training With Transvaginal Electrical Stimulation in Treating Female Stress Incontinence
Brief Title: A Comparison of Electrical Pudendal Nerve Stimulation and Pelvic Floor Muscle Training for Female Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZYSNXD-CC-ZDYJ010
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Stress Urinary Incontinence
Keywords: Electrical pudendal nerve stimulation; Pelvic floor muscle training; Transvaginal electrical stimulation; Stress urinary incontinence; Comparative study
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical pudendal nerve stimulation (Experimental): At a frequency of 2.5 Hz and an intensity (45~55 mA) as high as the patient can tolerate without discomfort; 60 minutes three times a week for a total of four weeks
  Interventions: Behavioral: Electrical pudendal nerve stimulation
- PFM training with Transvaginal ES (Active Comparator): PFM training: EMG-biofeedback assisted PFMT was performed by specially trained therapists, 20 min three times a week for a total of four weeks. Patients conduct 30 maximal high intensity PFM contractions for 2-6 sec (with 2-6 sec rest), three sessions a day at home for a total of four weeks.
  Transvaginal ES: At a current intensity of < 60 mA (as high as possible to get a contraction) and frequencies of 15 Hz and 85 Hz (alternate 3-min periods of stimulation); 20 min three times a week for a total of four weeks.
  Interventions: Behavioral: PFM training; Behavioral: Transvaginal ES

INTERVENTIONS:
Behavioral: Electrical pudendal nerve stimulation — Four sacral points are selected. The two upper points are located about 1 cm bilateral to the sacrococcygeal joint. On the upper points, a needle of 0.40 Х 100 mm is inserted perpendicularly to a depth of 80 to 90 mm to produce a sensation referred to the urethra or the anus. The locations of the two lower points are about 1 cm bilateral to the tip of the coccyx. On the lower points, a needle of 0.40 Х 100 or 125 mm is inserted obliquely towards the ischiorectal fossa to a depth of 90 to 110 mm to produce a sensation referred to the urethra. After the sensation referred to the above regions is produced, each of two pairs of electrodes from a G6805-2 Multi-Purpose Health Device is connected with the two ipsilaterally inserted needles.
  Arms: Electrical pudendal nerve stimulation
Behavioral: PFM training — A nerve function reconstruction treatment system (AM1000B; Shenzhen Creative Industry Co.Ltd, China) is used for EMG-biofeedback assisted PFMT.
  Arms: PFM training with Transvaginal ES
Behavioral: Transvaginal ES — A neuromuscular stimulation therapy system (PHENIX USB 4，Electronic Concept Lignon Innovation, France) is used for TES
  Arms: PFM training with Transvaginal ES

SUMMARY:
The purpose of this study is to determine whether electrical pudendal nerve stimulation is more effective than pelvic floor muscle training with Transvaginal electrical stimulation in treating female stress incontinence.

DETAILED DESCRIPTION:
Conservative therapy could be considered a choice of treatment for stress urinary incontinence (SUI) as it seems to have no side effects and causes significant and long-term improvement in symptoms. Pelvic floor muscle training (PFMT) and electrical stimulation are two commonly used forms of conservative treatment for SUI.

PFMT improves the structural support of the pelvis. However, many patients-especially women-have difficulty identifying and isolating their pelvic floor muscles (PFM) and are unable to perform the exercise effectively. Furthermore, patients who can identify the PFM often find that the required daily exercise routine is burdensome. Hence, the primary disadvantage of PFMT is lack of long-term patient compliance.

Electrical stimulation (ES) is a non-invasive, passive treatment that produces a muscle contraction. Transvaginal electrical stimulation (TES) has almost no side-effects and patient compliance in published reports is 70-85%. TES will result in PFM contraction by indirect nerve stimulation, mainly by polysynaptic reflex responses. The indirect stimulation and reflexive contraction may be the reason why the effect of electrical stimulation is not as good as that of PFMT when performed correctly.

By combining the advantages of PFMT and TES and incorporating the technique of deep insertion of long acupuncture needles, we developed electrical pudendal nerve stimulation (EPNS). In EPNS, long acupuncture needles of 0.40 Х 100 or 125 mm were deeply inserted into four sacral points and electrified to stimulate the pudendal nerves (PN) and contract the PFM. CT transverse plane at the coccygeal apex has showed that the position of the lower needle tip is similar to where (adjacent to PN at Alcock's canal) the Bion device is implanted for chronic PN stimulation. Besides the radiographic evidence, simultaneous records of perineal ultrasonographic PFM contraction, vaginal pressure and pelvic floor surface electromyogram in our previous study have proved that EPNS can exactly excite PN,contract the PFM and simulate PFMT. Our previous study has also proved that EPNS has a good therapeutic effect on female SUI. The purpose of this study is to compare the efficacy of EPNS to PFMT with TES in treating female SUI.

ELIGIBILITY:
Inclusion Criteria:

* SUI history
* Positive stress test result
* Urodynamically confirmed SUI
* Postvoid residual urine volume <50ml

Exclusion Criteria:

* Urge incontinence (overactive bladder or detrusor overactivity incontinence)
* Neurogenic bladder

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Stress test | 12 weeks

SECONDARY OUTCOMES:
A questionnaire to measure the severity of symptoms and the quality of life in SUI women | 12 weeks

OTHER OUTCOMES:
Pad test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, Master, Study Chair — Shanghai research institute of acupuncture and meridian
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

REFERENCES:
- [Background] Wang S, Zhang S. Simultaneous perineal ultrasound and vaginal pressure measurement prove the action of electrical pudendal nerve stimulation in treating female stress incontinence. BJU Int. 2012 Nov;110(9):1338-43. doi: 10.1111/j.1464-410X.2012.11029.x. Epub 2012 Mar 15. PMID 22417077
- [Derived] Wang S, Lv J, Feng X, Wang G, Lv T. Efficacy of Electrical Pudendal Nerve Stimulation in Treating Female Stress Incontinence. Urology. 2016 May;91:64-9. doi: 10.1016/j.urology.2016.02.027. Epub 2016 Feb 24. PMID 26921645